CLINICAL TRIAL: NCT03334630
Title: A Randomized Controlled Clinical Evaluation of the DiamondTemp™ Ablation System for the Treatment of Paroxysmal Atrial Fibrillation
Brief Title: DiamondTemp™ Ablation System for the Treatment of Paroxysmal Atrial Fibrillation
Acronym: DIAMOND-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TP00599
Record Dates: First submitted 2017-10-24; First posted 2017-11-07 (Actual); Results first posted 2020-12-09 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Paroxysmal Atrial Fibrillation; Atrial Fibrillation
Keywords: ablation; electrophysiology; atrial fibrillation; catheter; paroxysmal
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- DiamondTemp Ablation Catheter (Experimental): Catheter ablation to treat paroxysmal atrial fibrillation using DiamondTemp temperature-controlled ablation catheter
  Interventions: Device: DiamondTemp Ablation catheter
- TactiCath Quartz Ablation Catheter (Active Comparator): Catheter ablation to treat paroxysmal atrial fibrillation using TactiCath Quartz contact-force sensing ablation catheter
  Interventions: Device: TactiCath Quartz Ablation catheter

INTERVENTIONS:
Device: DiamondTemp Ablation catheter — a pulmonary vein isolation procedure will be performed using radiofrequency ablation catheter
  Arms: DiamondTemp Ablation Catheter
Device: TactiCath Quartz Ablation catheter — a pulmonary vein isolation procedure will be performed using radiofrequency ablation catheter
  Arms: TactiCath Quartz Ablation Catheter

SUMMARY:
The purpose of the DIAMOND-AF study is to establish the safety and effectiveness of the DiamondTemp System for the treatment of drug refractory, recurrent, symptomatic paroxysmal atrial fibrillation in patients.

DETAILED DESCRIPTION:
The DIAMOND-AF study is a prospective, single blind, 1:1 randomized controlled study being performed at multiple centers in the United States, Canada and Europe. The study will evaluate the safety and effectiveness of the DiamondTemp System used for ablation in patients with paroxysmal atrial fibrillation (AF). Subjects will be randomized for treatment with either the DiamondTemp Ablation Catheter or the TactiCath™ Quartz Contact Force Ablation Catheter manufactured by Abbott. Patients will be followed for 12 months.

ELIGIBILITY:
STUDY INCLUSION CRITERIA- Candidates must meet ALL the following criteria to be enrolled in the DIAMOND-AF study:

1. Above eighteen (18) years of age or of legal age to give informed consent specific to state and national law.
2. Subjects with a history of symptomatic, paroxysmal atrial fibrillation (PAF) who have had ≥2 episodes of PAF reported within the 6 months prior to index ablation procedure with a physician note indicating recurrent, self-terminating AF.
3. At least one episode of PAF documented by electrocardiographic data within the 12 months prior to index ablation procedure.
4. Refractory to at least one Class I-IV AAD for treatment of PAF.
5. Suitable candidate for intra-cardiac mapping and ablation of arrhythmia.
6. Subject agrees to comply with study procedures and be available (geographically stable) for follow-up visits for at least 12 months after enrollment.
7. Subject is willing and able to provide written consent.

STUDY EXCLUSION CRITERIA - Candidates will be excluded from the DIAMOND-AF study if any of the following conditions apply within the following timeframes:

At time of enrollment and/or prior to procedure:

1. AF secondary to electrolyte imbalance, thyroid disease or reversible or non-cardiac cause.
2. LA diameter > 5.5 cm.
3. LVEF < 35%.
4. Currently NYHA Class III or IV or exhibits uncontrolled heart failure.
5. BMI > 40 kg/m2.
6. LA ablation, septal closure device or mitral valve surgical procedure at any time prior to enrollment.
7. Presence of intramural thrombus, tumor or abnormality that precludes vascular access, catheter introduction or manipulation.
8. Coagulopathy, bleeding diathesis or suspected procoagulant state
9. Sepsis, active systemic infection or fever (>100.5°F / 38°C) within a week prior to the ablation procedure.
10. Significant restrictive or obstructive pulmonary disease or chronic respiratory condition.
11. Renal failure requiring dialysis or renal compromise that in the investigator's judgement would increase risk to the subject or deem the subject inappropriate to participate in the study.
12. Known allergies or intolerance to anticoagulant and antiplatelet therapies to be used in conjunction with the study or contrast sensitivity that cannot be adequately pre-treated prior to the ablation procedure.
13. Positive pregnancy test results for female subjects of childbearing potential or breast feeding.
14. Enrollment in a concurrent clinical study that in the judgement of the investigator would impact study outcomes.
15. Acute or chronic medical condition that in the judgment of the investigator would increase risk to the subject or deem the subject inappropriate to participate in the study.
16. Life expectancy < 12 months based on medical history or the medical judgement of the investigator.

    Within 1 month of enrollment or just prior to procedure:
17. Documented LA thrombus upon imaging.
18. Creatinine >2.5mg/dl or creatinine clearance <30mL/min.

    Within 2 months of enrollment:
19. Regularly (uninterrupted) prescribed amiodarone.

    Within 3 months of enrollment:
20. Significant GI bleed.
21. MI, unstable angina, cardiac surgery or coronary intervention.

    Within 6 months of enrollment:
22. CABG procedure.
23. ICD, CRT leads or pacemaker implant procedure.
24. Documented stroke, CVA, TIA or suspected neurological event.

    Within 12 months of enrollment:
25. An episode of AF lasting >7 days in duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josef Kautzner, MD, PhD, Principal Investigator — Institut klinické a experimentální medicíny (IKEM); William Maddox, MD, Principal Investigator — University of Alabama at Birmingham; Tom McElderry, MD, Principal Investigator — University of Alabama at Birmingham
Locations (23):
- United States (14):
  - Grandview Medical Center, Birmingham, Alabama
  - University Of Alabama, Birmingham, Alabama
  - Keck School Of Medicine, Los Angeles, California
  - Sequoia Hospital, Redwood City, California
  - Florida Hospital Orlando, Orlando, Florida
  - Ochsner Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Jackson Heart Clinic, Jackson, Mississippi
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, New York, New York
  - Trident Medical Center, Charleston, South Carolina
  - Medical University Of South Carolina, Charleston, South Carolina
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Houston Methodist Research Institute, Houston, Texas
- Southlake Regional Medical Centre, Toronto, Newmarket/Ontario, Canada
- Czechia (3):
  - Na Homolce, Prague, Prague
  - St Anne's University Hospital, Brno
  - Institut Klinicke a Experimentalni Mediciny (IKEM), Prague
- France (3):
  - Clinique Pasteur, Toulouse, Cedex 3
  - Clinique du Tonkin, Villeurbanne, Lyon
  - CHRU Nancy, Nancy
- Italy (2):
  - Centro Cardiologico Monzino, Milan, Milano
  - Ospedale dell'Angelo di Mestre, Mestre, Venezia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iwasawa J, Koruth JS, Petru J, Dujka L, Kralovec S, Mzourkova K, Dukkipati SR, Neuzil P, Reddy VY. Temperature-Controlled Radiofrequency Ablation for Pulmonary Vein Isolation in Patients With Atrial Fibrillation. J Am Coll Cardiol. 2017 Aug 1;70(5):542-553. doi: 10.1016/j.jacc.2017.06.008. PMID 28750697
- [Derived] Kautzner J, Albenque JP, Natale A, Maddox W, Cuoco F, Neuzil P, Poty H, Getman MK, Liu S, Starek Z, Dukkipati SR, Colley BJ 3rd, Al-Ahmad A, Sidney DS, McElderry HT. A Novel Temperature-Controlled Radiofrequency Catheter Ablation System Used to Treat Patients With Paroxysmal Atrial Fibrillation. JACC Clin Electrophysiol. 2021 Mar;7(3):352-363. doi: 10.1016/j.jacep.2020.11.009. Epub 2021 Jan 27. PMID 33516712

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment/randomization occurred between 06NOV2017 and 26OCT2018 across 23 sites in the US, Canada and Europe.
Groups:
- DiamondTemp Ablation Catheter: Catheter ablation to treat paroxysmal atrial fibrillation using the DiamondTemp temperature-controlled ablation catheter
  DiamondTemp Ablation catheter: a pulmonary vein isolation procedure will be performed using radiofrequency ablation catheter
- TactiCath Quartz Ablation Catheter: Catheter ablation to treat atrial fibrillation using the TactiCath Quartz contact-force sensing ablation catheter
  TactiCath Quartz Ablation catheter: a pulmonary vein isolation procedure will be performed using radiofrequency ablation catheter
Period: Overall Study
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Started | 239 | 243
Completed | 225 | 230
Not Completed | 14 | 13
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Lost to Follow-up | 3 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Enrollment closed | 2 | 1
Not completed — Subject not treated with study ablation due to technical difficulties | 0 | 1
Not completed — Subject unable to complete 12-month follow-up visit | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter | Total
Number analyzed (Participants) | 239 | 243 | 482
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (11.1) | 63.0 (10.4) | 62.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 100 | 203
  Male | 136 | 143 | 279
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 167 | 169 | 336
  Unknown or Not Reported | 66 | 69 | 135
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 159 | 161 | 320
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 73 | 74 | 147
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 0 | 1
  United States | 109 | 111 | 220
  Czechia | 61 | 62 | 123
  Italy | 2 | 3 | 5
  France | 66 | 67 | 133

OUTCOME MEASURES:

1. Primary Outcome: Safety: Freedom From a Composite of Pre-specified Serious Adverse Events (SAEs)
Description: The primary safety endpoint is defined as freedom from a composite of serious adverse events (SAE) occurring within 30-days and clinically symptomatic pulmonary vein stenosis through 6-months post-index ablation procedure, as adjudicated by an independent Clinical Events Committee (CEC) for relatedness to the procedure or device.
  The primary safety device- or procedure-related SAE composite will be the combined rate of the following events:
  * Atrioesophageal fistula
  * Bleeding complication
  * Cardiac tamponade / perforation
  * Death
  * Extended hospitalization
  * Myocardial infarction
  * Pericarditis
  * Phrenic nerve paralysis
  * Pulmonary edema
  * Pulmonary vein stenosis
  * Stroke post-ablation
  * Thromboembolism
  * Transient ischemic attack (TIA) post-ablation
  * Vagal nerve injury
  * Vascular access complications
Time Frame: Within 30-days or 6-months after index ablation procedure
Population: Intention-to-treat population: all randomized subjects are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 239 | 243
Participants
  Free from primary safety event | 231 | 227
  Not free from primary safety event | 8 | 16
Statistical Analysis 1: Comparison: DiamondTemp Ablation Catheter vs TactiCath Quartz Ablation Catheter; Null hypothesis: the DiamondTemp arm is inferior to the Control arm. Alternative hypothesis: the DiamondTemp arm is non-inferior to the Control arm; Test type: Non-Inferiority — Assuming a Control composite SAE freedom rate of 93.5%, 226 subjects per group yields 80% power to detect a non-inferiority margin of -6.5% between treatment groups at a significance level of 0.025; p < 0.0001, Farrington-Manning non-inferiority test — The a priori threshold for statistical significance is 0.025; Risk Difference (RD) = 0.0324, 95% CI 2-sided [-0.0132 to 0.0779] — Estimated risk difference = DiamondTemp composite SAE freedom rate - Control composite SAE freedom rate = 3.24% = 0.0324

2. Primary Outcome: Effectiveness: Freedom From Documented Atrial Fibrillation(AF), Atrial Flutter(AFL) and Atrial Tachycardia(AT) Episodes Following the Blanking Period (3M Post-ablation) Through the End of the Effectiveness Evaluation Period (12M Post-ablation).
Description: The primary effectiveness failure is defined by any of the following events:
  * Inability to electrically isolate all accessible targeted pulmonary veins during the ablation procedure
  * Documented episodes of AF, AFL or AT lasting ≥ 30 seconds in duration as evidenced by electrocardiographic data during the effectiveness evaluation period
  * DC cardioversion for AF, AFL or AT during the effectiveness evaluation period
  * A repeat ablation procedure to treat AF, AFL or AT during the effectiveness evaluation period
  * Use of a new or modification to existing Class I-IV anti-arrhythmic drug (AAD) regimen to treat AF, AFL or AT recurrence during the effectiveness evaluation period
  * Use of a non-study device for ablation of any AF targets during the index or repeat ablation procedure during the blanking period
  * More than one (1) repeat ablation procedure during the blanking period
Time Frame: 3-12M (3-12 months) after index ablation procedure
Population: Intention-to-treat population: all randomized subjects are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 239 | 243
Participants
  Free from primary effectiveness failure criteria | 189 | 184
  Not free from primary effectiveness failure criteria | 50 | 59
Statistical Analysis 1: Comparison: DiamondTemp Ablation Catheter vs TactiCath Quartz Ablation Catheter; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — Assuming a Control primary effectiveness rate of 65%, 229 subjects per group yields 80% power to detect a non-inferiority margin of -12.5% between treatment groups at a significance level of 0.025; p < 0.0001, Farrington-Manning non-inferiority test — The a priori threshold for statistical significance is 0.025; Risk Difference (RD) = 0.034, 95% CI 2-sided [-0.042 to 0.109] — Estimated risk difference = DiamondTemp composite SAE freedom rate - Control composite SAE freedom rate = 3.4% = 0.034

3. Secondary Outcome: Mean Duration of Individual Radiofrequency (RF) Ablations (Seconds)
Description: Mean duration of individual RF ablations (seconds) during the index ablation procedure
Time Frame: Index ablation procedure
Population: Subjects with measure available.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 235 | 238
seconds | 14.7 (5.3) | 32.6 (25.3)
Statistical Analysis 1: Comparison: DiamondTemp Ablation Catheter vs TactiCath Quartz Ablation Catheter; Null hypothesis: the population means for the DiamondTemp and Control groups are not different. Alternative hypothesis: the population means for the DiamondTemp and Control groups are different; Test type: Superiority — Four secondary endpoints will be tested for superiority over Control hierarchically with pre-specified order: 1. Mean duration of individual RF ablations (seconds) 2. Mean cumulative RF time per procedure (minutes) 3. Total fluoroscopy time (minutes) 4. Total procedure time (minutes) The first secondary endpoint needs to be significant at the two-sided 0.05 alpha level before the next one can be tested at the same threshold. Testing stops once an endpoint is determined to be non-significant; p < 0.0001, t-test, 2 sided — The a priori threshold for statistical significance is 0.05 two-sided. The p-value is adjusted for multiple comparisons via the hierarchical testing approach; Mean Difference (Final Values) = -17.9, 95% CI 2-sided [-21.2 to -14.6] — Difference is DiamondTemp minus Control. A lower value is better

4. Secondary Outcome: Mean Cumulative RF Time Per Procedure (Minutes)
Description: Mean cumulative RF time per procedure (minutes) during the index ablation procedure
Time Frame: Index ablation procedure
Population: Subjects with measure available.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 235 | 238
minutes | 17.9 (8.1) | 29.8 (14.0)
Statistical Analysis 1: Comparison: DiamondTemp Ablation Catheter vs TactiCath Quartz Ablation Catheter; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -11.9, 95% CI 2-sided [-13.9 to -9.8] — Difference is DiamondTemp minus Control. A lower value is better

5. Secondary Outcome: Freedom From a Composite of SAE Occurring Within 7-days
Description: Freedom from a composite of SAE occurring within 7-days post-index ablation procedure as adjudicated by an independent CEC for relatedness to the procedure or device.
  The device- or procedure-related SAE composite will be the combined rate of the following events:
  * Atrioesophageal fistula
  * Bleeding complication
  * Cardiac tamponade / perforation
  * Death
  * Extended hospitalization
  * Myocardial infarction
  * Pericarditis
  * Phrenic nerve paralysis
  * Pulmonary edema
  * Pulmonary vein stenosis
  * Stroke post-ablation
  * Thromboembolism
  * Transient ischemic attack (TIA) post-ablation
  * Vagal nerve injury
  * Vascular access complications
Time Frame: Within 7-days after the index ablation procedure
Population: Intention-to-treat population: all randomized subjects are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 239 | 243
Participants
  Free from composite SAEs within 7 days | 231 | 230
  Not free from composite SAEs within 7 days | 8 | 13

6. Secondary Outcome: Freedom From Documented AF, AT and AFL Episodes in the Absence of Class I and III Anti-arrhythmic Drugs (AADs).
Description: Freedom from documented AF, AT and AFL episodes following the blanking period through 12-month follow-up post-ablation procedure in the absence of class I and III anti-arrhythmic drug therapy.
Time Frame: 3-12 months after index ablation procedure
Population: Intention-to-treat population: all randomized subjects are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 239 | 243
Participants
  Free from documented AF, AT and AFL episodes in the absence of class I and III AADs | 142 | 120
  Not free from documented AF, AT and AFL episodes in the absence of class I and III AADs | 97 | 123

7. Secondary Outcome: Rate of Acute Procedural Success
Description: Rate of acute procedural success is defined as confirmation of electrical isolation of PVs via assessment of entrance block at least 20 minutes following the last ablation around the respective PV.
Time Frame: Index ablation procedure
Population: Intention-to-treat population: all randomized subjects are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 239 | 243
Participants
  Acute procedural success | 228 | 228
  Not acute procedural success | 11 | 15

8. Secondary Outcome: Rate of Single Procedure Success With Freedom From Documented AF, AT and AFL at 12 Months.
Description: Rate of single procedure success is defined as the rate of subjects treated with one single ablation procedure during study participation and with freedom from documented AF, AT and AFL at 12 months.
Time Frame: Index ablation procedure through 12-months after index ablation procedure
Population: Intention-to-treat population: all randomized subjects are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 239 | 243
Participants
  Single procedure success | 183 | 185
  Not single procedure success | 56 | 58

9. Secondary Outcome: Rate of Single Procedure Success With Freedom From ALL Primary Effectiveness Endpoint Failure Criteria.
Description: Rate of single procedure success is defined as the rate of subjects treated with one single ablation procedure during study participation and with freedom from ALL primary effectiveness endpoint failure criteria.
Time Frame: Index ablation procedure through 12-months after index ablation procedure
Population: Intention-to-treat population: all randomized subjects are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 239 | 243
Participants
  Single procedure success | 175 | 173
  Not single procedure success | 64 | 70

10. Secondary Outcome: Rate of Occurrence of Electrically Reconnected Pulmonary Veins (PVs)
Description: Rate of occurrence of electrically reconnected PVs following a 20-minute waiting period assessed by entrance block at index procedure.
Time Frame: Index ablation procedure
Population: Intention-to-treat population: all randomized subjects are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 239 | 243
Participants
  Occurrence of electrically reconnected PVs | 45 | 45
  No occurrence of electrically reconnected PVs | 194 | 198

11. Secondary Outcome: Accumulated Changes in Quality of Life (QOL) Using the Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) Questionnaire
Description: Accumulated changes in QOL using the AF QOL Survey (AFEQT Questionnaire) from baseline through 6 and 12 months following ablation procedure.
  The Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) Questionnaire is an atrial fibrillation-specific health-related quality of life Questionnaire. The overall AFEQT score can range from 0 to 100, with 0 corresponding to complete disability and 100 corresponding to no disability. So a higher AFEQT score means a better outcome.
Time Frame: Baseline, 6-months after index ablation and 12-months after index ablation
Population: Subjects with measure available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 215 | 219
score on a scale
  Change from baseline to 6 months: number analyzed (Participants) | 207 | 209
  Change from baseline to 6 months | 27.8 (23.1) | 25.5 (22.7)
  Change from baseline to 12 months | 31.1 (23.4) | 30.1 (23.2)

12. Secondary Outcome: Neurological Changes Measured Using the National Institutes of Health Stroke Scale (NIHSS)
Description: Neurological changes measured using the NIH stroke scale between baseline and post-ablation (pre-discharge visit) and at 12 months post-ablation procedure.
  The National Institutes of Health Stroke Scale (NIHSS) is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. The total NIHSS score can range from 0 to 42, with 0 indicating no stroke symptoms and 42 indicating extremely severe stroke symptoms. So a higher NIHSS score means a worse outcome.
Time Frame: Baseline, pre-discharge after index ablation and 12-months after index ablation procedure
Population: Subjects with measure available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 216 | 222
score on a scale
  Change from baseline to 6 months | 0 (0.30) | 0 (0.32)
  Change from baseline to 12 months: number analyzed (Participants) | 214 | 212
  Change from baseline to 12 months | -0.1 (0.36) | -0.1 (0.38)

13. Secondary Outcome: Total Procedure Time (Minutes)
Description: Total procedure time (minutes) at index procedure is defined as time of first assigned ablation catheter insertion into the vasculature to time of last procedural ablation catheter removed.
Time Frame: Index ablation procedure
Population: Subjects with measure available.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 235 | 240
minutes | 109.7 (46.2) | 115.4 (50.8)
Statistical Analysis 1: Comparison: DiamondTemp Ablation Catheter vs TactiCath Quartz Ablation Catheter; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; [p-value comment as in outcome 3, analysis 1]; Since the previous secondary endpoint (Total fluoroscopy time) was non-significant, testing stopped and this secondary endpoint was not tested; Mean Difference (Final Values) = -5.7, 95% CI 2-sided [-14.4 to 3.1] — Difference is DiamondTemp minus Control. A lower value is better

14. Secondary Outcome: Time to Achieve Initial Pulmonary Vein Isolation (PVI) (Minutes)
Description: Time to achieve initial PVI (minutes) at index procedure is defined as time of delivery of first RF ablation with the assigned ablation catheter until confirmation of PVI.
Time Frame: Index ablation procedure
Population: Subjects with measure available.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 235 | 238
minutes | 65.7 (29.9) | 69.4 (35.2)

15. Secondary Outcome: Total Treatment Device Time (Minutes)
Description: Total treatment device time (minutes) at index procedure is defined as time of delivery of first RF ablation with the assigned ablation treatment catheter to removal of the treatment catheter.
Time Frame: Index ablation procedure
Population: Subjects with measure available.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 235 | 239
minutes | 83.1 (34.0) | 91.4 (60.9)

16. Secondary Outcome: Total Number of RF Ablations Per Procedure
Description: Total number of RF ablations per procedure at index procedure
Time Frame: Index ablation procedure
Population: Subjects with measure available.
Measure: Mean (Standard Deviation); unit: counts
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 232 | 238
counts | 74.2 (32.9) | 71.1 (39.8)

17. Secondary Outcome: Total Fluid Infused Through the Ablation Catheter (mL)
Description: Total fluid infused through the assigned ablation catheter (mL) at index procedure
Time Frame: Index ablation procedure
Population: Subjects with measure available.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 235 | 237
mL | 332.2 (120.8) | 785.2 (351.5)

18. Secondary Outcome: Total Fluoroscopy Time (Minutes)
Description: Total fluoroscopy time (minutes) at index procedure
Time Frame: Index ablation procedure
Population: Subjects with measure available.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 232 | 239
minutes | 12.7 (10.2) | 12.8 (9.4)
Statistical Analysis 1: Comparison: DiamondTemp Ablation Catheter vs TactiCath Quartz Ablation Catheter; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.8528, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.9 to 1.6] — Difference is DiamondTemp minus Control. A lower value is better

19. Secondary Outcome: Number of Re-hospitalizations Due to Atrial Fibrillation Recurrence After Blanking Period
Description: Number of re-hospitalizations due to atrial fibrillation recurrence after blanking period
Time Frame: 3-12 months after index ablation procedure
Population: Intention-to-treat population: all randomized subjects are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
Number analyzed (Participants) | 239 | 243
Participants
  0 re-hospitalization | 221 | 229
  1 re-hospitalization | 17 | 13
  2 re-hospitalizations | 1 | 1

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) observed by the Investigator or staff during a physical or laboratory examination, interventional procedure or mentioned by the subject, either spontaneously or upon questioning, were recorded on an AE case report form, from the time of signed informed consent through the twelve-month follow-up visit.
Arm/Group | DiamondTemp Ablation Catheter | TactiCath Quartz Ablation Catheter
All-Cause Mortality (participants affected / at risk) | 0/239 | 0/243
Serious Adverse Events (participants affected / at risk) | 34/239 | 43/243
Other Adverse Events (participants affected / at risk) | 32/239 | 41/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DiamondTemp Ablation Catheter (N=239) | TactiCath Quartz Ablation Catheter (N=243)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 10 (14) | 3 (3)
Atrial flutter (Cardiac disorders) | 2 (2) | 6 (6)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac perforation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Colonic abscess (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Cranial nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Venous injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemochromatosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
IVth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Phrenic nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Seizure like phenomena (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 1 (1)
Device pacing issue (Product Issues) | 0 (0) | 1 (1)
Renal disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Arthrodesis (Surgical and medical procedures) | 1 (1) | 0 (0)
Colostomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DiamondTemp Ablation Catheter (N=239) | TactiCath Quartz Ablation Catheter (N=243)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Atrial flutter (Cardiac disorders) | 4 (4) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 3 (3)
Pericarditis (Cardiac disorders) | 3 (3) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 3 (3)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 4 (4)
Chest pain (General disorders) | 3 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (5)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 6 (6) | 3 (3)
Headache (Nervous system disorders) | 4 (4) | 3 (3)
Syncope (Nervous system disorders) | 3 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Haematoma (Vascular disorders) | 1 (1) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
While the language in each agreement may vary slightly, in general it states that the Principal Investigator (PI) agrees to not independently discuss/publish trial results until a multi-center publication is released. If the multi-center publication is not submitted within one year after study completion across all centers, PIs may publish the results pertaining to their activities. PI must submit this request to the Sponsor for review/comment at least forty-five (45) days prior to submission.

DOCUMENTS (8):
  • Study Protocol: Revision I (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT03334630/Prot_001.pdf
  • Study Protocol: Revision G (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT03334630/Prot_002.pdf
  • Study Protocol: Revision F (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT03334630/Prot_003.pdf
  • Study Protocol: Revision E (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT03334630/Prot_004.pdf
  • Study Protocol: Revision D (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT03334630/Prot_005.pdf
  • Study Protocol: Revision C (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/30/NCT03334630/Prot_006.pdf
  • Study Protocol: Revision H (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT03334630/Prot_007.pdf
  • Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT03334630/SAP_000.pdf